CLINICAL TRIAL: NCT00407160
Title: Comparison of Two Different Immunosuppression Protocols in Highly Sensitized Renal Transplant Recipients: Campath Induction With Tacrolimus Monotherapy vs Thymoglobulin Induction With Triple Drug Protocol.
Brief Title: A Trial of Tolerogenic Immunosuppression in Highly Sensitized Renal Transplant Recipients
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 04-245
Record Dates: First submitted 2006-11-21; First posted 2006-12-04 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2012-12

CONDITIONS: Kidney Diseases
Keywords: Kidney transplant; Tolerance induction; High Panel Reactive Antibody (PRA) kidney recipients
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1 Standard Immunosuppression: Anti-thymocyte Globulin (Rabbit)] ,tacrolimus, mycophenolate mofetil and prednisone
  Patients with End Stage Renal Disease (ESRD) and high Panel Reactive Antibody (PRA) who randomize to the control group. These patients will get induction therapy prior to transplant with Thymoglobulin 1.5 mg/kg/day for 4 days to a total dose of 6mg/kg.
  They will receive maintenance immunosuppression with three drugs : tacrolimus, cellcept and prednisone.
- Group 2 Campath Immunosuppression: Alemtuzumab,tacrolimus
  Patients with ESRD and high PRA who randomize to the study group. These patients will get induction therapy prior to reperfusion of the kidney, during the transplant operation, with Campath (Alemtuzumab) 30mg, one dose. They will receive maintenance immunosuppression with tacrolimus alone (monotherapy).

SUMMARY:
Comparison between Campath induction and monotherapy with Tacrolimus vs Thymoglobulin induction and triple drug maintenance using Tacrolimus, mycophenolate, and steroids.

DETAILED DESCRIPTION:
Recent reports suggest that it might be possible to induce a state of tolerance in solid organ transplantation. So called "tolerogenic immunosuppression" involves induction with lymphocyte depleting antibodies followed by monotherapy with calcineurin inhibitors, cyclosporin or tacrolimus. The proposed study aims to evaluate a protocol of immunosuppression induction with lymphocyte depleting antibody Campath given prior to graft reperfusion, followed by tacrolimus monotherapy in highly sensitized patients (PRA >14% or past historical =/>50% and/or multiple renal transplants) undergoing renal transplantation, and compare it with the current standard protocol at UTMB which employs induction with Thymoglobulin given over 4 days followed by 3 drugs: tacrolimus, mycophenolate and steroids. In both groups of patients the target tacrolimus levels will be the same i.e, between 10 to 15ng/mL, soon after the transplant. In the Campath gro up, tacrolimus will be tapered after 3 months in patients who do not have rejection and appear to be developing donor specific tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18-75 years.
2. Recipients of multiple kidney transplants
3. Patients with a PRA >14% and/or a past historical PRA greater or equal to 50%.
4. Females of childbearing potential must have a negative pregnancy test prior to inclusion.
5. Patients who are willing and able to participate in the full course of the study and from whom written informed consent has been obtained.

Exclusion Criteria:

1. Patients with a history of malignancy within the last 5 years, except excised squamous or basal cell carcinoma of the skin.
2. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after contraception and until the termination of gestation,confirmed by a positive human chorionic gonadotropin(hCG) laboratory test.
3. Patients who are HIV positive.
4. Patients with symptoms of significant somatic or mental illness or evidence of current drug and/or alcohol abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end stage renal disease , on dialysis, who are regarded as "high immunological risk" becuase they have lost previous transplants to rejection, or have a high panel reactive antibody (PRA).
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2004-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
graft survival | 1 year
  Cumulative graft survival at 1 year

SECONDARY OUTCOMES:
rejection episodes | 1 year
  1 year cumulative freedom from rejection

CONTACTS AND LOCATIONS:
Overall Officials: Philip G Thomas, MD, Principal Investigator — UTMB Department of Surgery
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Background] Calne RY. Prope tolerance: a step in the search for tolerance in the clinic. World J Surg. 2000 Jul;24(7):793-6. doi: 10.1007/s002680010127. PMID 10833245
- [Background] Magliocca JF, Knechtle SJ. The evolving role of alemtuzumab (Campath-1H) for immunosuppressive therapy in organ transplantation. Transpl Int. 2006 Sep;19(9):705-14. doi: 10.1111/j.1432-2277.2006.00343.x. PMID 16918530
- [Derived] Thomas PG, Woodside KJ, Lappin JA, Vaidya S, Rajaraman S, Gugliuzza KK. Alemtuzumab (Campath 1H) induction with tacrolimus monotherapy is safe for high immunological risk renal transplantation. Transplantation. 2007 Jun 15;83(11):1509-12. doi: 10.1097/01.tp.0000263344.53000.a1. PMID 17565326